CLINICAL TRIAL: NCT04834921
Title: Randomized Blinded Controlled Pilot Study on Clinical Assessment of Continuous Hemodialysis With a High Molecular Flux Membrane
Brief Title: MCO Membrane Efficiency in Septic Shock Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fiorenza Ferrari (Other)
Collaborators: International Renal Research Institute Vicenza (Other); University of Giessen (Other)
Responsible Party: Sponsor-Investigator, Fiorenza Ferrari, Senior Consultant at intensive Care Unit of Hospital San Matteo, Pavoa, Italy, Fondazione IRCCS Policlinico San Matteo di Pavia
Organization: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 46/15A
Record Dates: First submitted 2021-03-30; First posted 2021-04-08 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: Septic Shock; Acute Kidney Injury
Keywords: Renal Replacement Therapy,; Cytokines; Efficiency
MeSH Terms: conditions — Shock, Septic; Acute Kidney Injury

STUDY DESIGN:
Intervention Model Description: All patients received two consecutive RRT (MCO-CVVHD and HFF-CVVHDF); in a controlled randomized (1:1) blinded manner. Each RRT treatment lasted 24 hours Crossover randomized to sequence (A+B or B+A) for 48 h total without washout
Who Masked: Investigator
Masking Description: Blinding procedure was limited to the doctors who collected the data and the external statistician who performed the analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MCO-CVVHD (Experimental): CVVHD with MCO filter for 24 hours
  Interventions: Device: Ultraflux® EMiC®2
- HFF-CVVHDF (Active Comparator): CVVHDF with high flux filter for 24 hours
  Interventions: Device: Ultraflux® EMiC®2

INTERVENTIONS:
Device: Ultraflux® EMiC®2 — Ultraflux® EMiC®2-CVVHD runs in septic shock patients with AKI KDIGO 3 for 24 hours. and patients were randomised to start Ultraflux® EMiC®2-CVVHD in the first day or in the second day from the RRT start; more precisely, crossover randomized to sequence consists in Ultraflux® EMiC®2-CVVHD (first day)+ HFF-CVVHDF(second day) and HFF-CVVHDF (first day) + Ultraflux® EMiC®2-CVVHD (second day) for 48 h total without washout
  Other Names: HFF-CVVHDF

SUMMARY:
This is a monocentre randomized pilot study. All patients received two consecutive RRT: CVVHD with MCO filter (Ultraflux® EMiC®2) and post-Continuous Veno-Venous Hemodiafiltration (CVVHDF) with HFF(AV1000S®) in a controlled randomized (1:1) blinded manner. Crossover randomized to sequence (A+B or B+A) for 48 h total without washout.

DETAILED DESCRIPTION:
This is a monocentre randomized pilot study. All patients received CVVHD with MCO filter (Ultraflux® EMiC®2) and post-Continuous Veno-Venous Hemodiafiltration (CVVHDF) with HFF(AV1000S®) in a controlled randomized (1:1) blinded manner. Crossover randomized to sequence (A+B or B+A) for 48 h total without washout.

The efficiency of the filters for small and middle molecules was compared in septic shock patients with AKI stage 3.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years;
* septic shock according to ACCP/SCCM criteria
* AKI KDIGO stage 3
* clinical decision to begin citrate based-RRT for at least 48 hours
* Hb >= 9 g/dL
* Obtain the informed consent

Exclusion Criteria:

* Pre-existing chronic renal insufficiency
* Weight > 125 kg Life expectancy <24 hr
* Declared do Not Resuscitate or Comfort Measures
* Platelets < 20 [10^3/ul] or active bleeding
* Pregnancy
* Contraindication to citrate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-12-31 (Actual); Primary Completion 2020-02-21 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
improvement in haemodynamic parameters | 48 hours
  measurements of the hemodynamic parameters: mean arterial pressure (MAP, mmHg)
improvement in haemodynamic parameters | 48 hours
  measurements of the hemodynamic parameters: heart rate (HR, beat/min)
improvement in haemodynamic parameters | 48 hours
  measurements of the hemodynamic parameters: lactate level (mmol/L)
improvement in haemodynamic parameters | 48 hours
  measurements of the hemodynamic parameters: cardiac index (CI; L/min/m2)
improvement in haemodynamic parameters | 48 hours
  measurements of the hemodynamic parameters: stroke volume variation (SVV; %)
improvement in haemodynamic parameters | 48 hours
  measurements of the hemodynamic parameters: PVC (mmHg)
improvement in haemodynamic parameters | 48 hours
  measurements of the hemodynamic parameters: SVRI (dyn*s/cm5*m2)
improvement in haemodynamic parameters | 48 hours
  measurements of the hemodynamic parameters: SCVO2 (%)
improvement in haemodynamic parameters | 48 hours
  measurements of the hemodynamic parameters: dose of vasopressor or inotropes (mcg/kg/min)

SECONDARY OUTCOMES:
clerance of cytokine | 48 hours
  removal of IL-6 (pg/mL)
clerance of cytokine | 48 hours
  removal of IL-10 (pg/mL); reduction was evaluated after before and after the RRT
clerance of cytokine | 48 hours
  removal of IL-8 (pg/mL); reduction was evaluated after before and after the RRT
clerance of cytokine | 48 hours
  removal of MPO (U/L); reduction was evaluated after before and after the RRT
Efficiency for middle molecules | 48 hours
  measure of the efficacy (Kcd, (ml/kg/h)) of removal of B2microglobulin for each filter according to equation in Neri M, Villa G, Garzotto F, Bagshaw S, Bellomo R, Cerda J, Ferrari F, Guggia S, Joannidis M, Kellum J, Kim JC, Mehta RL, Ricci Z, Trevisani A, Marafon S, Clark WR, Vincent JL, Ronco C; Nomenclature Standardization Initiative (NSI) alliance. Nomenclature for renal replacement therapy in acute kidney injury: basic principles. Crit Care. 2016 Oct 10;20(1):318. Review.
Efficiency for small molecules | 48 hours
  measure of the efficacy (Kcd (ml/kg/h)) of BUN for each filter according to equation in Neri M, Villa G, Garzotto F, Bagshaw S, Bellomo R, Cerda J, Ferrari F, Guggia S, Joannidis M, Kellum J, Kim JC, Mehta RL, Ricci Z, Trevisani A, Marafon S, Clark WR, Vincent JL, Ronco C; Nomenclature Standardization Initiative (NSI) alliance. Nomenclature for renal replacement therapy in acute kidney injury: basic principles. Crit Care. 2016 Oct 10;20(1):318. Review.
Efficiency for small molecules | 48 hours
  measure of Efficacy (Kcd Cr (ml/kg/h)) of removal of SCr for each filter according to equation in Neri M, Villa G, Garzotto F, Bagshaw S, Bellomo R, Cerda J, Ferrari F, Guggia S, Joannidis M, Kellum J, Kim JC, Mehta RL, Ricci Z, Trevisani A, Marafon S, Clark WR, Vincent JL, Ronco C; Nomenclature Standardization Initiative (NSI) alliance. Nomenclature for renal replacement therapy in acute kidney injury: basic principles. Crit Care. 2016 Oct 10;20(1):318. Review.
removal of antibiotics | 48 hours
  evaluation of plasma level of vancomycin piperacillin/tazobactam(mcg/ml)
removal of antibiotics | 48 hours
  evaluation of plasma level of vancomycin (mcg/ml)
removal of antibiotics | 48 hours
  evaluation of plasma level of meropenem(mg/L)

CONTACTS AND LOCATIONS:
Locations (1):
- Fiorenza Ferrari, Pavia, PV, Italy

IPD SHARING:
Plan to Share IPD: No